CLINICAL TRIAL: NCT05102227
Title: Cardiac ResynchronizatiOn and arrhythmiaS Sensing Via the LEFT Bundle. The CROSS LEFT Study.
Brief Title: Cardiac ResynchronizatiOn and arrhythmiaS Sensing Via the LEFT Bundle.
Acronym: CROSS LEFT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Principal Investigator, Nicolas Clementy, MD, PhD, Associate Professor, University Hospital, Tours
Other Study IDs: CROSS LEFT
Record Dates: First submitted 2021-10-04; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Left Bundle Branch Area Pacing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LBBAP: Patients implanted with a dual-chamber DF-1 cardioverter-defibrillator. Ventricular tachy sensing is performed via an IS-1 pacing lead placed in the interventricular septum.
  Interventions: Device: Left bundle branch area pacing

INTERVENTIONS:
Device: Left bundle branch area pacing — A dual-chamber DF-1 defibrillator is implanted. Left bundle branch area pacing is performed for cardiac resynchronization therapy.
  Other Names: Cardioverter-defibrillator implantation

SUMMARY:
Evaluation of ventricular arrhythmias sensing via a left bundle branch area pacing lead.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or non-ischemic cardiomyopathy
* Left ventricular ejection fraction ≤35% despite optimal medical therapy
* Left bundle branch block with QRS ≥130 milliseconds

Exclusion Criteria:

* Previously implanted intra-cardiac material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with an indication of a new implantation of a cardiac resynchronization therapy system.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful defibrillation at 35 Joules. | 24 hours
  After manual induction of ventricular fibrillation, a 35 Joules will be delivered with the implanted defibrillator.

SECONDARY OUTCOMES:
Time from ventricular fibrillation induction to defibrillation shock. | 24 hours
  After manual induction of ventricular fibrillation, the duration of appropriate ventricular sensing will be measured until the 35 Joules shock is delivered.
Number of appropriate and inappropriate arrhythmic episodes. | 6 months
  The occurrence of appropriately or inappropriately detected episodes with a high ventricular rate ≥170 beats-per-minute will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Tours, Tours, Please Select..., France

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared with manuscript reviewers, upon reasonable request.

REFERENCES:
- [Derived] Clementy N, Bodin A, Ah-Fat V, Babuty D, Bisson A. Dual-chamber ICD for left bundle branch area pacing: the cardiac resynchronization and arrhythmia sensing via the left bundle (cross-left) pilot study. J Interv Card Electrophysiol. 2023 Jun;66(4):905-912. doi: 10.1007/s10840-022-01342-6. Epub 2022 Aug 16. PMID 35970951